CLINICAL TRIAL: NCT04062188
Title: Development and Validation of the Telephone Interview Form for Stroke Outcome
Brief Title: VAlidity and Reliability of the Telephone Interview Form for Stroke Outcome Evaluation
Acronym: ARISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, President of Institute for Brain Disorders, Beijing University of Chinese Medicine, Dongzhimen Hospital, Beijing
Other Study IDs: 2018-JYBZZ-XS147
Record Dates: First submitted 2019-08-15; First posted 2019-08-20 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Stroke
Keywords: Stroke outcomes; Telephone interview; Modified Rankin Scale questionnaire; Barthel Index questionnaire; Validity study; Reliability study
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Telephone Interview Form — Telephone Interview Form is an original simple questionnaire developed based on the combination of Barthel Index questionnaire and simplified modified Rankin Scale questionnaire with internal rules.
  Other Names: Telephone Interview Questionnaire

SUMMARY:
The investigators combined the mRS questionnaire and BI questionnaire and then developed a telephone interview form as a simple questionnaire with internal rules. The main purpose of this study is to evaluate the validity and reliability of the telephone interview form when compared with face-to-face assessment in clinically stable patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of ischemic or hemorrhagic stroke.
* The course of 1 to 12 months.
* Patient or procuratorial caregiver has a good understanding so as to answer rater's telephone interview.
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Patients with psychological or mental disorders.
* Patients suffer from other so severe diseases that they can't complete the follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population are clinically stable stroke patients with the course between 1 to 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-12-22 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Criterion validity of the Telephone Interview Form | Baseline, 3 days after baseline, 6 days after baseline
  The agreement between the Telephone Interview Form and face-to-face assessment.
Inter-rater reliability of the Telephone Interview Form | 3 days after baseline, 6 days after baseline
  The agreement of the Telephone Interview Form when administrated by two different rates

SECONDARY OUTCOMES:
Sensitivity of Telephone Interview Form | 3 days after baseline, 6 days after baseline
  Sensitivity of Telephone Interview Form when administered by telephone compared with face-to-face at various cut-off values
Specificity of Telephone Interview Form | 3 days after baseline, 6 days after baseline
  Specificity of Telephone Interview Form when administered by telephone compared with face-to-face at various cut-off values
Internal consistency reliability of Barthel Index questionaire in Telephone Interview Form | Baseline, 3 days after baseline, 6 days after baseline
  Internal consistency reliability of Barthel Index questionaire will be evaluated.
Convergent validity of Telephone Interview Form | Baseline, 3 days after baseline, 6 days after baseline
  Relationship between Telephone Interview Form and other scales (i.e. (National Institute of Health stroke scale)

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, Principal Investigator — Dongzhimen Hospital affiliated to Beijing University of Chinese
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided